CLINICAL TRIAL: NCT06495762
Title: Preventing Premature Family Maladjustment: an e-Health Interdisciplinary Research
Acronym: e-ParWelB
Status: Not yet recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: Catholic University of the Sacred Heart (Other); Treviso Regional Hospital (Network); Ospedale San Bortolo di Vicenza (Other); Azienda Ospedaliero Universitaria di Cagliari (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); IRCCS Ospedale San Raffaele (Other); Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Alessandra Decataldo, Senior Associate Professor, University of Milano Bicocca
Other Study IDs: 20225R7XB3
Record Dates: First submitted 2024-06-24; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Psychological Distress
Keywords: Preterm birth; Parental well-being; Sociology of Health; Digital-Based Monitoring; Mixed-method Research; e-Health
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: e-health assesment — This study is purely observational and does not forsee any intervention but only observational assesment of parents' wellbeing

SUMMARY:
The consequences of preterm birth extend beyond the clinical conditions of the newborn, profoundly impacting the functioning and well-being of families. Although various research examines changes in parents' well-being and perception of self-efficacy during the stay in NICU, there is a lack of research analyzing what happens in the delicate transition phase at home after the baby's discharge. Recently, scholars have advocated for the use of web-based and app-based support programs both to monitor and prevent preterm family maladjustment and to assist parents struggling with the transition home. The main aim of this interdisciplinary research project is to develop a socio-psychological model focused on assessing the well-being of parents of premature infants during and after their stay in a NICU. Specifically, the study aims to (1) monitor the mental health of parents of premature infants, both at the time of the child's discharge from the NICU and in the first six months after discharge to prevent family maladjustment, (2) deepen our understanding of the role of digital tools in monitoring and supporting the well-being of parents of premature infants, and (3) study the potential impact of the relationship with healthcare professionals on the overall well-being of parents. The project combines mixed methods of social research and psychological support with an e-health approach. The well-being of parents of premature infants will be assessed using validated scales administered through a questionnaire to parents of preterm infants within six NICUs at the time of the child's discharge. Subsequently, a follow-up assessment of parental well-being will be implemented through the administration of the validated scales in a web app. Additionally, an ethnographic phase will be conducted in the NICUs, involving observation of the interaction between healthcare professionals and parents, as well as narrative interviews with healthcare staff. It is expected to shed light on the determinants of well-being among parents of premature infants, in relation to varying levels of prematurity severity, socio-demographic characteristics such as gender, age, and socioeconomic status, and parental involvement in NICU care practices. With the follow-up phase via web app, the project also aims to prevent family maladjustment by providing psychological support and utilizing an e-health tool.

DETAILED DESCRIPTION:
Brief statement of primary study objectives and the main secondary study objectives.

The e-ParWelB project is an interdisciplinary study which, starting from the premises of the ParWelB project, aims to evaluate the well-being of preterm parents during and after hospitalization in the Neonatal Intensive Care Unit NICU using research strategies such as standardized questionnaires with internationally validated scales and psychological support with an innovative and technology-driven approach. Recently scholars have supported the use of Web-App-based support programs to monitor and prevent maladjustment of preterm families and assist parents who have difficulty transitioning from the NICU to home (Sawyer et al., 2019; Greene et al., 2020). Furthermore, the work of Garfield et al. (2016) with very low birth weight infants demonstrated that parents who received an app-based support program improved self-efficacy and their perception of preparedness for discharge.

Starting from these premises, the main objectives of our research can be summarised as follows: (1) monitor the mental health of parents of children born prematurely, with a six-month follow-up to prevent family maladjustment ; (2) deepen knowledge on the role of digital tools in monitoring and supporting the mental health of parents whose infants have been admitted to neonatal intensive care for critical health situations such as prematurity.

Brief statement of primary study outcome and primary estimand/estimator. Then describe the main secondary study outcome measures.

Considering the time and economic resources available, we estimate to intercept the families of approximately 175 children born preterm, thus roughly a sample of 350 participants.

The validated scales employed will be used to create statistical indices measuring concepts such as levels of stress, depression, parental self-efficacy and perception of social support received from parents. These variables will be correlated through statistical processing and modelling with independent socio-demographic variables (gender, age, nationality, ...), and indicators of economic, social and cultural capital.

The research assumes to find statistically significant differences in the levels of stress, anxiety and self-efficacy with respect to sample segmentations related to gender, educational background and migration variables.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children born before 36+6 of gestational age (GA).
* The parents must be at least 18 years old
* Children must have been hospitalized in intensive or sub-intensive care for at least ten days.
* Parents must be able to speak fluent Italian or English.

Exclusion Criteria:

- Children must not have other genetic pathologies or other pathologies not linked to the preterm birth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents of preterm child who were born in one of the partner NICU during the monitoring phase of the project.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-09-02 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Anxiety | The scale is administered 3 times: the day of child discharge from NICU (starting from 01/09/2024 to 28/02/2025), 30 days after child's discharge (from 01/10/2024 to 28/03/2025) and 180 days after child's discharge (from 01/03/2024 to 28/09/2025).
  Measured through Postpartum Specific Anxiety Scale (PSAS). Most of the literature on postpartum anxiety (Glasheen, Richardson, & Fabio, 2010; Lostein, 2007; Meades & Ayers, 2011) refers to measures of generalised anxiety which can often prove problematic from a psychometric point of view. To date, the only questionnaire available that specifically measures postpartum anxiety is the Postpartum Specific Anxiety Scale (PSAS). The instrument also demonstrated excellent psychometric properties (ω between 0.72 and 0.90 in the four scales and λ4 between 0.71 and 0.92 in the four scales). For these reasons, the research team believed it was the most sensitive and suitable tool for capturing the construct under investigation in the target population (parents of children born preterm).
Post-partum PTSD | The scale is administered 2 times: the day of child discharge from NICU (starting from 01/09/2024 to 28/02/2025) and 90 days after child's discharge (from 01/12/2024 to 28/05/2025).
  Measured through City Birth Trauma Scale (City BiTS). The scale is an instrument specifically developed to measure birth-related post-traumatic stress disorder according to the recent DSM-5 criteria and is, to the authors' knowledge, the only instrument with this specificity. This instrument has previously demonstrated excellent reliability (Cronbach's a = 0.92). For these reasons, the research team believed it was the most sensitive and suitable tool for capturing the construct under investigation in the target population (parents of children born preterm).
Post-partum depression | The scale is administered 2 times: the day of child discharge from NICU (starting from 01/09/2024 to 28/02/2025) and 90 days after child's discharge (from 01/12/2024 to 28/05/2025).
  Measured through Edinbugh Postnatal Depression Scale (EPDS). Postnatal depression is the most widely measured disorder in the postpartum population which in Italy is mostly subject to routine checks. The Edinburgh Postnatal Depression Scale (EPDS) is the most widely used self-report questionnaire to measure postpartum depression given the simplicity of administration, ease of cultural adaptation and excellent psychometric properties demonstrated. The validated Italian version demonstrated good validity and reliability (Cronbach's α =0.7894), confirming the validity of the EPDS in identifying postnatal depression.
Post-partum parent-child bonding | The scale is administered once, the day of child discharge from NICU (starting from 01/09/2024 to 28/02/2025).
  Measured through Postpartum Bonding Questionnaire (PBQ) (in T0). The scale aims to measure the quality of the bond between parents and children and identify if there are problems in the relationship. The Italian adaptation of the PBQ, edited by Rosario Montirosso, Claudia Fedeli, Livio Provenzi and Ian Brockington was developed using the back-translation procedure (Montirosso et al., 2009). Studies show that the Italian version of the PBQ has good psychometric properties and can be implemented in the Italian cultural context to assess early mother-child relational difficulties (Busonera et al., 2017).
Parenting-related stress | The scale is administered 3 times: 30 days after child's discharge from NICU (from 01/10/2024 to 28/03/2025), 60 days after child's discharge from NICU (from 01/11/2024 to 28/04/2025) and 180 days after child's discharge (from 01/03/2024 to 28/09/2025).
  Measured through Parenting Stress Index (PSI). The literature on existing research has highlighted the possibility of identifying stressful "child-parent" systems early in order to develop interventions aimed at reducing stress that can reduce the frequency and the intensity of emotional and behavioral disorders of children in our society (Cash et al., 2006; van Ijzendoorn et al., 2005). The Parenting Stress Index (PSI) was developed in response to the need for a measure to assess these characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Decataldo, PhD, Principal Investigator — University of Milano Bicocca
Locations (6):
- Italy (6):
  - Dipartimento Materno infantile, Terapia Intensiva Neonatale, Azienda Ospedaliero-Universitaria di Cagliari, Cagliari, CA
  - S.C. Neonatologia e Terapia Intensiva Neonatale, I.R.C.C.S. Ospedale San Gerardo Monza, Monza, MB
  - U.O Neonatologia e Patologia Neonatale, I.R.C.C.S. Ospedale San Raffaele, Milan, MI
  - S.C. Neonatologia e Terapia Intensiva Neonatale, Fondazione IRCCS Policlinico San Matteo di Pavia., Pavia, PV
  - U.O.C. di Terapia Intensiva Neonatale, patologia neonatale ed assistenza al neonato sano presso il Presidio Ospedaliero di Treviso, Treviso, TV
  - UOSD di Terapia Intensiva e Patologia Neonatale presso l'ospedale di Vicenza (ULSS 8 Berica)., Vicenza, VI

IPD SHARING:
Plan to Share IPD: No